CLINICAL TRIAL: NCT03191799
Title: A Single-Arm, Multicenter Phase IIIB Clinical Trial to Evaluate the Safety and Tolerability of Prophylactic Emicizumab in Hemophilia A Patients With Inhibitors
Brief Title: A Study to Evaluate the Safety and Tolerability of Prophylactic Emicizumab in Hemophilia A Patients With Inhibitors
Acronym: STASEY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO39129; 2016-004366-25 (EudraCT Number)
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Results first posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1.5 mg/kg Emicizumab QW (Experimental): Participants will receive initial weekly doses of prophylactic emicizumab subcutaneously for 4 weeks, followed by maintenance doses consisting of half the initial dose, administered subcutaneously for the remainder of the 2-year treatment period
  Interventions: Drug: Emicizumab

INTERVENTIONS:
Drug: Emicizumab — Initial dosing will be 3 mg/kg/week subcutaneously for 4 weeks; Maintenance dosing will follow at 1.5 mg/kg/week subcutaneously for the remainder of the 2-year treatment period
  Other Names: Hemlibra; RO5534262; ACE910

SUMMARY:
This is a phase IIIb, single arm, open-label, multi-center study to evaluate the safety and tolerability of emicizumab in participants with congenital hemophilia A who have documented inhibitors against Factor VIII (FVIII) at enrollment. Approximately 200 participants, aged 12 or older, will be enrolled in this study and are expected to be enrolled at approximately 85 sites globally. Participants will receive an initial weekly dose of prophylactic emicizumab subcutaneously for 4 weeks, followed by a weekly maintenance dose subcutaneously for the remainder of the 2-year treatment period.

ELIGIBILITY:
Inclusion Criteria:

* As per investigator's judgement, a willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures, including the patient-reported outcome (PRO) questionnaires and bleed diaries through the use of an electronic device or paper
* Aged 12 years or older at the time of informed consent
* Diagnosis of congenital hemophilia A with persistent inhibitors against FVIII
* Documented treatment with bypassing agents or FVIII concentrates in the last 6 months (on-demand or prophylaxis). Prophylaxis needs to be discontinued the latest by a day before starting emicizumab
* Adequate hematologic, hepatic, and renal function
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a highly effective contraceptive method with a failure rate of <1% per year during the treatment period and for at least five elimination half-lives (24 weeks) after the last dose of emicizumab

Exclusion Criteria:

* Inherited or acquired bleeding disorder other than hemophilia A
* Ongoing (or plan to receive during the study) immune tolerance induction (ITI) therapy (prophylaxis regimens with FVIII and/or bypassing agents must be discontinued prior to enrollment). Patients receiving ITI therapy will be eligible following the completion of a 72-hour washout period prior to the first emicizumab administration
* History of illicit drug or alcohol abuse within 12 months prior to screening, as per the investigator's judgment
* High risk for thrombotic microangiopathy (TMA) (e.g., have a previous medical or family history of TMA), as per the investigator's judgment
* Previous (in the past 12 months) or current treatment for thromboembolic disease (with the exception of previous catheter-associated thrombosis for which antithrombotic treatment is not currently ongoing) or current signs of thromboembolic disease
* Other conditions (e.g., certain autoimmune diseases) that may increase the risk of bleeding or thrombosis
* History of clinically significant hypersensitivity reaction associated with monoclonal antibody therapies or components of the emicizumab injection
* Known human immunodeficiency virus (HIV) infection with CD4 count <200 cells/μL within 6 months prior to screening
* Use of systemic immunomodulators (e.g., interferon or rituximab) at enrollment or planned use during the study, with the exception of antiretroviral therapy
* Concurrent disease, treatment, or abnormality in clinical laboratory tests that could interfere with the conduct of the study or that would, in the opinion of the investigator or Sponsor, preclude the patient's safe participation in and completion of the study or interpretation of the study results
* Receipt of: Emicizumab in a prior investigational study; An investigational drug to treat or reduce the risk of hemophilic bleeds within five half-lives of last drug administration; A non-hemophilia-related investigational drug within last 30 days or five half-lives, whichever is shorter; or, Any concurrent investigational drug.
* Pregnancy or lactation, or intent to become pregnant during the study
* Positive serum pregnancy test result within 7 days prior to initiation of emicizumab (females only)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (72):
- Australia (3):
  - Royal Prince Alfred Hospital; Haematology, Camperdown, New South Wales
  - Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- UZ Leuven Gasthuisberg, Leuven, Belgium
- Brazil (4):
  - Centro de Hematologia E Hemoterapia Do Parana - Hemepar, Curitiba, Paraná
  - Instituto Estadual de Hema, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clinicas - UNICAMP, Campinas, São Paulo
  - Faculdade de Medicina de Ribeirão Preto - Universidade de Sao Paulo, Ribeirão Preto, São Paulo
- Canada (4):
  - Kaye Edmonton Clinic, Edmonton, Alberta
  - CancerCare Manitoba; Neuro-Oncology, Winnipeg, Manitoba
  - McMaster University Health Sciences Center, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
- Colombia (2):
  - Centro de Atención e Investigación Médica CAIMED S.A.S, Localidad Puente Aranda
  - Hospital Pablo Tobon Uribe, Medellín
- Helsingin yliopistollinen keskussairaala, Meilahden sairaala, Helsinki, Finland
- Germany (6):
  - Vivantes Klinikum im Friedrichshain - Landsberger Allee, Angiologie und Hämostaseologie, Berlin
  - Universitätsklinikum Bonn; Institut für Experimentelle Hämatologie und Transfusionsmedizin, Bonn
  - Hämophiliezentrum Med. Klinik III/Institut für Transfusionsmedizin; Johann Wolfgang Goethe-Univers., Frankfurt/M.
  - Universitätsklinikum Leipzig, Innere Medizin, Neurologie, Dermatologie; Zentrum für Hämostaseologie, Leipzig
  - Hämophilie-Zentrum Rhein Main GmbH, Mörfelden-Walldorf
  - Klinikum der Universität München, Campus Innenstadt; Hämostaseologische Ambulanz/Hämophiliezentrum, München
- Oncomedica, Guatemala City, Guatemala
- Hungary (3):
  - Magyar Honvédség Egészségügyi Központ; Országos Haemophilia Központ, Budapest
  - Országos Vérellátó Szolgálat - Győri Regionális Vérellátó Központ, Győr
  - University of Pecs, I st Dept of Internal Medicine, Pécs
- India (7):
  - St. John's Medical College & Hospital; Department of Medicine, Bengaluru, Karnataka
  - King Edward Memorial Hospital and Seth G.S. Medical College; Department of Hematology, Mumbai, Maharashtra
  - Fortis Hospitals Limited, Mumbai, Maharashtra
  - Sahyadri Speciality Hospital; Hematology & Bone Marrow Unit, Pune, Maharashtra
  - Christian Medical College & Hospital; Department of Haematology, Vellore, Maharashtra
  - Nil Ratan Sircar Medical College and Hospital; Department of Hematology, Kolkata, West Bengal
  - Grant Medical Foundation, Ruby Hall Clinic, Pune
- Sheba Medical Center - National Hemophilia Center, Tel Litwinsky, Israel
- Italy (9):
  - AOU Federico II; Medicina Clinica Chirurgia Centro Emocoaugulopatie e Emofilia, Napoli, Campania
  - AOU Policlinico S. Orsola Malpighi; U.O. Angiologia e Malattie della Coagulazione Marino Golinelli, Bologna, Emilia-Romagna
  - AOU di Parma; Dip Emergenza-Urgenza Centro Riferimento Regionale per l'emofilia, Parma, Emilia-Romagna
  - Universita' Degli Studi La Sapienza-Ist.Di Ematologia; Dip Biot Cel e Ematol, Rome, Lazio
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico; Centro Emofilia e Trombosi "Angelo Bianchi e Bonomi", Milan, Lombardy
  - AO Città Salute e Scienza D-Osp S. G. Battista Molinette; SSCVD Malattie Tromboti e Emorragiche, Turin, Piedmont
  - Azienda Uni Ria Policlinico P. Giaccone ; Divisione Di Ematologia E Trapianto, Palermo, Sicily
  - AOU Careggi; SOD Malattie Emorragiche, Florence, Tuscany
  - Azienda Ospedaliera di Padova; Centro Emofilia, Padua, Veneto
- Mexico (3):
  - Hospital General de México, Distrito Federal, Mexico CITY (federal District)
  - CENTRO MEDICO NACIONAL SIGLO XXI; Banco de Sangre, Mexico City, Mexico CITY (federal District)
  - Hospital de Especialidades Centro Medico Nacional La Raza; Haematology, Mexico City
- Netherlands (2):
  - Erasmus MC / location Sophia Kinderziekenhuis, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Complejo Hospitalario Arnulfo Arias Madrid; Servicio de Hematología, Panama City, Panama
- Instytut Hematologii i Transfuzjologii; Klinika Zaburzeń Hemostazy i Chorób Wewnętrznych, Warsaw, Poland
- Portugal (3):
  - Hospital Geral; Servico de Imuno-Hemoterapia, Coimbra
  - Hospital de Santa Maria; Servico de Imuno-Hemoterapia; Servico de Imuno-Hemoterapia, Lisbon
  - Hospital de Sao Joao; Servico de Imuno-Hemoterapia; Servico de Imuno-Hemoterapia, Porto
- Louis Turcanu Emergency Clinical Hospital for Children; First Pediatric Clinic, Timișoara, Romania
- Russia (5):
  - Regional State Budgetary Institution of Healthcare "Regional Cinilcal Hospital"; Pulmonology, Barnaul, Altayskiy Kray
  - Morozov Children's Municipal Clinical Hospital. Haematology department, Moscow
  - "Hematological Scientific Center, Moscow
  - City Outpatient Clinic #37, City Hemophilia Treatment Center, Saint Petersburg
  - Samara State Medical University, Samara
- King Faisal Specialist Hospital & Research Centre; Oncology, Riyadh, Saudi Arabia
- Spain (5):
  - Hospital Universitario Vall de Hebron; Unidad de Hemofília, Barcelona
  - Hospital Universitario la Paz; Servicio de Hematologia, Madrid
  - Hospital Regional Universitario Carlos Haya; Servicio de Hematologia, Málaga
  - Hospital Universitario Virgen del Rocio; Servicio de Hematologia, Seville
  - Hospital Universitario la Fe; Servicio de Hematologia, Valencia
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset; Koagulationscentrum, Gothenburg
  - Karolinska Universitetssjukhuset; Koagulationsmottagningen, Solna
- Inselspital Bern; Hämatologie und Hämatologisches Zentrallabor, Bern, Switzerland
- United Kingdom (5):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - The Royal London Hospital, London
  - Royal Free Hospital, London
  - Royal Victoria Infirmary; Non-Malignant Haematology Research, Newcastle upon Tyne
  - Royal Hallamshire Hospital Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

REFERENCES:
- [Derived] Castaman G, Peyvandi F, Kremer Hovinga JA, Schutgens REG, Robson S, Moreno K, Jimenez-Yuste V. Surgical Experience from the STASEY Study of Emicizumab Prophylaxis in People with Hemophilia A with Factor VIII Inhibitors. TH Open. 2024 Jan 12;8(1):e42-e54. doi: 10.1055/s-0043-1777766. eCollection 2024 Jan. PMID 38222041

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 195 patients were enrolled in the clinical trial.
Groups:
- 1.5 mg/kg Emicizumab QW: Participants were enrolled to receive initial weekly doses of prophylactic 3.0 mg/kg emicizumab subcutaneously (SC) for 4 weeks, followed by prophylactic maintenance doses consisting of 1.5 mg/kg emicizumab once a week (QW), administered SC for the remainder of the 2-year treatment period.
Period: Overall Study
Arm/Group | 1.5 mg/kg Emicizumab QW
Started (Intent-to-Treat (ITT) Population) | 195
Received at Least One Dose of Emicizumab (Safety Population) | 193
Dose Up-Titrated to 3 mg/kg QW | 2
Completed | 186
Not Completed | 9
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 1
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 195
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.2 (16.6)
Age, Customized [Count of Participants; unit: Participants]
  ≥12 to <18 Years Old | 40
  ≥18 to <65 Years Old | 146
  ≥65 Years Old | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41
  Not Hispanic or Latino | 143
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 19
  Asian | 38
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 121
  More than one race | 0
  Unknown or Not Reported | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Summary of the Number of Participants With Adverse Events, Severity Assessed According to the World Health Organization (WHO) Toxicity Grading Scale
Description: Investigators sought information on adverse events (AEs) at each contact with participants. The WHO toxicity grading scale was used for assessing AE severity (i.e., intensity of an AE); any AEs not specifically listed in the WHO toxicity grading scale were assessed for severity according to the following grades: Grade 1 is mild; Grade 2 is moderate, Grade 3 is severe; Grade 4 is life-threatening; and Grade 5 is death. Regardless of severity, some AEs may have also met seriousness criteria. The terms "severe" and "serious" are not synonymous; severity and seriousness were independently assessed for each AE. aPCC = activated prothrombin complex concentrate
Time Frame: From Baseline until study completion (up to 2 years)
Population: Safety Population: all participants who received at least one dose of emicizumab
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 193
Participants
  Any Adverse Event (AE) | 163
  Fatal AE | 2
  Serious AE | 31
  AE Leading to Withdrawal from Treatment | 1
  AE Leading to Dose Modification/Interruption | 4
  AE Leading to Study Discontinuation | 1
  Grade 3-5 AE | 39
  Related AE | 35
  Local Injection Site Reaction | 22
  Systemic Hypersensitivity/Anaphylac(tic/toid) Reaction | 0
  Thromboembolic Event (TE) | 2
  TE Related to aPCC and Emicizumab | 0
  Thrombotic Microangiopathy (TMA) | 0
  TMA Related to aPCC and Emicizumab | 0
  Cases of Potential Drug-Induced Liver Injury | 0
  Suspected Transmission of Infectious Agent by the Study Drug | 0

2. Primary Outcome: Adverse Events (AEs) Rates Per 100 Patient-Years for All-Grade AEs, Serious AEs, and Grade ≥3 AEs
Description: Investigators sought information on adverse events (AEs) at each contact with participants. The WHO toxicity grading scale was used for assessing AE severity (i.e., intensity of an AE); any AEs not specifically listed in the WHO toxicity grading scale were assessed for severity according to the following grades: Grade 1 is mild; Grade 2 is moderate, Grade 3 is severe; Grade 4 is life-threatening; and Grade 5 is death. Regardless of severity, some AEs may have also met seriousness criteria. The terms "severe" and "serious" are not synonymous; severity and seriousness were independently assessed for each AE. The AE rate per 100 patient-years was computed as follows: AE Rate = (Number of AEs observed/ Total patient-years at risk)*100. Total patient-years at risk is the sum over all patients of the time intervals (in years) between start of study therapy (study day 1) and the end of follow up.
Time Frame: From Baseline until study completion (up to 2 years)
Population: Safety Population: all participants who received at least one dose of emicizumab
Measure: Number (95% Confidence Interval); unit: AEs per 100 patient-years
Units Other Than Participants: Adverse Events (AEs)
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 193
Number analyzed (Adverse Events (AEs)) | 800
AEs per 100 patient-years
  All-Grade AEs | 211.92 [197.49 to 227.13]
  Serious AEs: number analyzed (Adverse Events (AEs)) | 50
  Serious AEs | 13.25 [9.83 to 17.46]
  Grade ≥3 AEs: number analyzed (Adverse Events (AEs)) | 65
  Grade ≥3 AEs | 17.22 [13.29 to 21.95]

3. Primary Outcome: Number of Participants by Hematology and Biochemistry Laboratory Parameter Test Results as Shifts From the WHO Toxicity Grade at Baseline to the Worst WHO Toxicity Grade Post-Baseline
Description: The World Health Organization (WHO) toxicity grading scale was used for determining the severity of laboratory abnormalities (i.e., test results outside of the reference range) for hematology and biochemistry parameters; Grade 0 is normal and Grades 1 to 4 represent worsening levels of the parameter outside of the normal range in the specified direction of the abnormality (high and low are above and below the range, respectively). Not every laboratory abnormality qualified as an adverse event (AE). A laboratory test result was reported as an AE if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment; resulted in a medical intervention or a change in concomitant therapy; or was clinically significant in the investigator's judgment. Baseline was defined as the last available assessment prior to first receipt of study drug. Abs = absolute count; SGOT/AST = aspartate aminotransferase; SGPT/ALT = alanine aminotransferase
Time Frame: Baseline, Weeks 2, 3, and 5; Months 3, 6, 9, 12, and 18; and at Early Termination/Study Completion (up to 24 months)
Population: Safety Population: all participants who received at least one dose of emicizumab
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 193
Participants
  Hemoglobin, Low - Grade 0 to 0 | 173
  Hemoglobin, Low - Grade 0 to 1 | 8
  Hemoglobin, Low - Grade 0 to 2 | 4
  Hemoglobin, Low - Grade 0 to 4 | 1
  Hemoglobin, Low - Grade 1 to 0 | 1
  Hemoglobin, Low - Grade 1 to 1 | 2
  Hemoglobin, Low - Grade 1 to 2 | 1
  Hemoglobin, Low - Grade 1 to 3 | 1
  Hemoglobin, Low - Grade 2 to 1 | 1
  Hemoglobin, Low - Grade 2 to 3 | 1
  Neutrophils, Total (Abs), Low - Grade 0 to 0 | 173
  Neutrophils, Total (Abs), Low - Grade 0 to 1 | 13
  Neutrophils, Total (Abs), Low - Grade 0 to 2 | 1
  Neutrophils, Total (Abs), Low - Grade 0 to 3 | 2
  Neutrophils, Total (Abs), Low - Grade 0 to 4 | 2
  Neutrophils, Total (Abs), Low - Grade 1 to 1 | 2
  Platelets, Low - Grade 0 to 0 | 190
  Platelets, Low - Grade 0 to 1 | 2
  Platelets, Low - Grade 1 to 0 | 1
  Alkaline Phosphatase, High - Grade 0 to 0 | 187
  Alkaline Phosphatase, High - Grade 0 to 1 | 3
  Alkaline Phosphatase, High - Grade 0 to 2 | 1
  Alkaline Phosphatase, High - Grade 1 to 1 | 2
  Bilirubin, High - Grade 0 to 0 | 169
  Bilirubin, High - Grade 0 to 1 | 14
  Bilirubin, High - Grade 1 to 0 | 3
  Bilirubin, High - Grade 1 to 1 | 2
  Bilirubin, High - Grade 1 to 2 | 3
  Bilirubin, High - Grade 2 to 2 | 2
  Blood Urea Nitrogen, High - Grade 0 to 0 | 187
  Blood Urea Nitrogen, High - Grade 0 to 1 | 5
  Blood Urea Nitrogen, High - Grade 1 to 1 | 1
  Calcium (Corrected), High - Grade 0 to 0 | 192
  Calcium (Corrected), High - Grade 1 to 2 | 1
  Calcium (Corrected), Low - Grade 0 to 0 | 173
  Calcium (Corrected), Low - Grade 0 to 1 | 15
  Calcium (Corrected), Low - Grade 0 to 2 | 1
  Calcium (Corrected), Low - Grade 1 to 0 | 3
  Calcium (Corrected), Low - Grade 1 to 1 | 1
  Creatinine, High - Grade 0 to 0 | 185
  Creatinine, High - Grade 0 to 1 | 5
  Creatinine, High - Grade 0 to 2 | 1
  Creatinine, High - Grade 1 to 1 | 1
  Creatinine, High - Grade 1 to 2 | 1
  Glucose, High - Grade 0 to 0 | 148
  Glucose, High - Grade 0 to 1 | 28
  Glucose, High - Grade 0 to 2 | 6
  Glucose, High - Grade 1 to 1 | 2
  Glucose, High - Grade 1 to 2 | 3
  Glucose, High - Grade 2 to 2 | 1
  Glucose, High - Grade 2 to 3 | 1
  Glucose, High - Grade 3 to 2 | 1
  Glucose, High - Grade 3 to 3 | 2
  Glucose, High - Grade 4 to 3 | 1
  Glucose, Low - Grade 0 to 0 | 180
  Glucose, Low - Grade 0 to 1 | 7
  Glucose, Low - Grade 0 to 2 | 4
  Glucose, Low - Grade 1 to 0 | 2
  Magnesium, Low - Grade 0 to 0 | 188
  Magnesium, Low - Grade 0 to 1 | 4
  Magnesium, Low - Grade 1 to 1 | 1
  Phosphorus, Low - Grade 0 to 0 | 160
  Phosphorus, Low - Grade 0 to 1 | 21
  Phosphorus, Low - Grade 1 to 0 | 2
  Phosphorus, Low - Grade 1 to 1 | 9
  Phosphorus, Low - Grade 1 to 2 | 1
  Potassium, High - Grade 0 to 0 | 189
  Potassium, High - Grade 0 to 1 | 2
  Potassium, High - Grade 0 to 2 | 1
  Potassium, High - Grade 0 to 4 | 1
  Potassium, Low - Grade 0 to 0 | 184
  Potassium, Low - Grade 0 to 1 | 6
  Potassium, Low - Grade 1 to 0 | 3
  SGOT/AST, High - Grade 0 to 0 | 164
  SGOT/AST, High - Grade 0 to 1 | 13
  SGOT/AST, High - Grade 0 to 2 | 8
  SGOT/AST, High - Grade 1 to 0 | 1
  SGOT/AST, High - Grade 1 to 1 | 5
  SGOT/AST, High - Grade 1 to 2 | 1
  SGOT/AST, High - Grade 1 to 3 | 1
  SGPT/ALT, High - Grade 0 to 0 | 158
  SGPT/ALT, High - Grade 0 to 1 | 22
  SGPT/ALT, High - Grade 0 to 2 | 5
  SGPT/ALT, High - Grade 1 to 0 | 1
  SGPT/ALT, High - Grade 1 to 1 | 4
  SGPT/ALT, High - Grade 1 to 2 | 2
  SGPT/ALT, High - Grade 1 to 4 | 1
  Sodium, High - Grade 0 to 0 | 178
  Sodium, High - Grade 0 to 1 | 7
  Sodium, High - Grade 0 to 2 | 2
  Sodium, High - Grade 1 to 0 | 4
  Sodium, High - Grade 1 to 1 | 2
  Sodium, Low - Grade 0 to 0 | 166
  Sodium, Low - Grade 0 to 1 | 19
  Sodium, Low - Grade 0 to 2 | 2
  Sodium, Low - Grade 1 to 0 | 3
  Sodium, Low - Grade 1 to 1 | 2
  Sodium, Low - Grade 1 to 2 | 1

4. Primary Outcome: Change From Baseline in Body Temperature at Specified Timepoints
Description: Vital signs that were measured included body temperature, pulse and respiratory rates, systolic and diastolic blood pressure, and weight. On treatment days, measurement occurred prior to emicizumab administration.
Time Frame: Baseline, Weeks 2, 3, and 5; Months 3, 6, 9, 12, and 18; and at Early Termination/Study Completion (up to 24 months)
Population: Safety Population: all participants who received at least one dose of emicizumab. The number analyzed included participants with a baseline value and a post-baseline value at a given timepoint.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 193
degrees Celsius
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 192
  Baseline (BL) - Value at Visit | 36.33 (0.52)
  Change from BL at Week 2: number analyzed (Participants) | 190
  Change from BL at Week 2 | 0.04 (0.41)
  Change from BL at Week 3: number analyzed (Participants) | 191
  Change from BL at Week 3 | 0.03 (0.40)
  Change from BL at Week 5: number analyzed (Participants) | 191
  Change from BL at Week 5 | 0.03 (0.45)
  Change from BL at Month 3: number analyzed (Participants) | 187
  Change from BL at Month 3 | 0.04 (0.45)
  Change from BL at Month 6: number analyzed (Participants) | 183
  Change from BL at Month 6 | 0.07 (0.50)
  Change from BL at Month 9: number analyzed (Participants) | 184
  Change from BL at Month 9 | 0.06 (0.48)
  Change from BL at Month 12: number analyzed (Participants) | 182
  Change from BL at Month 12 | 0.07 (0.48)
  Change from BL at Month 18: number analyzed (Participants) | 176
  Change from BL at Month 18 | 0.10 (0.53)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 163
  Change from BL at Early Termination/Study Completion | 0.08 (0.48)

5. Primary Outcome: Change From Baseline in Systolic Blood Pressure at Specified Timepoints
Description: as for outcome 4
Time Frame: Baseline, Weeks 2, 3, and 5; Months 3, 6, 9, 12, and 18; and at Early Termination/Study Completion (up to 24 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimetres of mercury (mmHg)
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 193
millimetres of mercury (mmHg)
  Baseline (BL) - Value at Visit | 121.1 (14.3)
  Change from BL at Week 2 | -0.9 (11.1)
  Change from BL at Week 3: number analyzed (Participants) | 192
  Change from BL at Week 3 | -1.2 (10.6)
  Change from BL at Week 5: number analyzed (Participants) | 192
  Change from BL at Week 5 | -1.3 (12.3)
  Change from BL at Month 3: number analyzed (Participants) | 188
  Change from BL at Month 3 | 0.1 (11.5)
  Change from BL at Month 6: number analyzed (Participants) | 185
  Change from BL at Month 6 | -0.2 (13.1)
  Change from BL at Month 9: number analyzed (Participants) | 186
  Change from BL at Month 9 | 0.1 (13.1)
  Change from BL at Month 12: number analyzed (Participants) | 184
  Change from BL at Month 12 | 0.1 (13.9)
  Change from BL at Month 18: number analyzed (Participants) | 177
  Change from BL at Month 18 | -0.1 (13.8)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 166
  Change from BL at Early Termination/Study Completion | 1.9 (14.1)

6. Primary Outcome: Change From Baseline in Diastolic Blood Pressure at Specified Timepoints
Description: as for outcome 4
Time Frame: Baseline, Weeks 2, 3, and 5; Months 3, 6, 9, 12, and 18; and at Early Termination/Study Completion (up to 24 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimetres of mercury (mmHg)
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 193
millimetres of mercury (mmHg)
  Baseline (BL) - Value at Visit | 75.5 (10.4)
  Change from BL at Week 2 | -1.2 (8.5)
  Change from BL at Week 3: number analyzed (Participants) | 192
  Change from BL at Week 3 | -1.0 (8.9)
  Change from BL at Week 5: number analyzed (Participants) | 192
  Change from BL at Week 5 | -1.2 (9.2)
  Change from BL at Month 3: number analyzed (Participants) | 188
  Change from BL at Month 3 | -0.3 (9.8)
  Change from BL at Month 6: number analyzed (Participants) | 185
  Change from BL at Month 6 | -0.7 (10.1)
  Change from BL at Month 9: number analyzed (Participants) | 186
  Change from BL at Month 9 | -1.3 (9.4)
  Change from BL at Month 12: number analyzed (Participants) | 184
  Change from BL at Month 12 | -1.2 (10.4)
  Change from BL at Month 18: number analyzed (Participants) | 177
  Change from BL at Month 18 | -0.9 (9.6)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 166
  Change from BL at Early Termination/Study Completion | 0.0 (11.0)

7. Primary Outcome: Change From Baseline in Pulse Rate at Specified Timepoints
Description: as for outcome 4
Time Frame: Baseline, Weeks 2, 3, and 5; Months 3, 6, 9, 12, and 18; and at Early Termination/Study Completion (up to 24 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 193
beats per minute
  Baseline (BL) - Value at Visit | 76.6 (11.6)
  Change from BL at Week 2 | 1.0 (9.9)
  Change from BL at Week 3: number analyzed (Participants) | 192
  Change from BL at Week 3 | 1.6 (11.6)
  Change from BL at Week 5: number analyzed (Participants) | 192
  Change from BL at Week 5 | -0.5 (11.3)
  Change from BL at Month 3: number analyzed (Participants) | 188
  Change from BL at Month 3 | -0.8 (10.4)
  Change from BL at Month 6: number analyzed (Participants) | 185
  Change from BL at Month 6 | -0.7 (11.6)
  Change from BL at Month 9: number analyzed (Participants) | 186
  Change from BL at Month 9 | -1.0 (11.3)
  Change from BL at Month 12: number analyzed (Participants) | 184
  Change from BL at Month 12 | -0.5 (12.2)
  Change from BL at Month 18: number analyzed (Participants) | 177
  Change from BL at Month 18 | -2.1 (12.7)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 166
  Change from BL at Early Termination/Study Completion | -1.2 (11.9)

8. Primary Outcome: Change From Baseline in Respiratory Rate at Specified Timepoints
Description: as for outcome 4
Time Frame: Baseline, Weeks 2, 3, and 5; Months 3, 6, 9, 12, and 18; and at Early Termination/Study Completion (up to 24 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 193
breaths per minute
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 192
  Baseline (BL) - Value at Visit | 17.0 (3.1)
  Change from BL at Week 2: number analyzed (Participants) | 192
  Change from BL at Week 2 | 0.2 (2.2)
  Change from BL at Week 3: number analyzed (Participants) | 191
  Change from BL at Week 3 | 0.0 (2.3)
  Change from BL at Week 5: number analyzed (Participants) | 189
  Change from BL at Week 5 | -0.1 (2.5)
  Change from BL at Month 3: number analyzed (Participants) | 187
  Change from BL at Month 3 | 0.3 (4.7)
  Change from BL at Month 6: number analyzed (Participants) | 180
  Change from BL at Month 6 | -0.1 (2.5)
  Change from BL at Month 9: number analyzed (Participants) | 184
  Change from BL at Month 9 | 0.0 (2.7)
  Change from BL at Month 12: number analyzed (Participants) | 180
  Change from BL at Month 12 | 0.3 (2.9)
  Change from BL at Month 18: number analyzed (Participants) | 173
  Change from BL at Month 18 | -0.4 (2.7)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 160
  Change from BL at Early Termination/Study Completion | -0.7 (3.1)

9. Primary Outcome: Change From Baseline in Body Weight at Specified Timepoints
Description: as for outcome 4
Time Frame: Baseline, Weeks 2, 3, and 5; Months 3, 6, 9, 12, and 18; and at Early Termination/Study Completion (up to 24 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 193
kilograms (kg)
  Baseline (BL) - Value at Visit | 69.55 (16.60)
  Change from BL at Week 2 | 0.14 (1.06)
  Change from BL at Week 3: number analyzed (Participants) | 192
  Change from BL at Week 3 | 0.34 (1.18)
  Change from BL at Week 5: number analyzed (Participants) | 192
  Change from BL at Week 5 | 0.52 (1.56)
  Change from BL at Month 3: number analyzed (Participants) | 188
  Change from BL at Month 3 | 0.98 (2.44)
  Change from BL at Month 6: number analyzed (Participants) | 186
  Change from BL at Month 6 | 1.11 (3.20)
  Change from BL at Month 9: number analyzed (Participants) | 186
  Change from BL at Month 9 | 1.61 (4.08)
  Change from BL at Month 12: number analyzed (Participants) | 184
  Change from BL at Month 12 | 1.85 (4.88)
  Change from BL at Month 18: number analyzed (Participants) | 177
  Change from BL at Month 18 | 2.58 (5.56)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 165
  Change from BL at Early Termination/Study Completion | 3.15 (6.78)

10. Secondary Outcome: Model-Based Annualized Bleed Rates (ABR) for Treated Bleeds, All Bleeds, Treated Joint Bleeds, Treated Target Joint Bleeds, and Treated Spontaneous Bleeds
Description: The number of bleeds over the efficacy period was analyzed as an ABR using a negative binomial regression model. Treated bleeds: bleeds followed by a hemophilia medication reported to be a "Treatment for bleed". All bleeds: included both treated and non-treated bleeds. Treated joint bleeds: treated bleeds where bleed type was "joint bleed" accompanied by at least one of following symptoms: "increased swelling or warmth of the skin over the joint", "increasing pain" or "decreased range of motion or difficulty using the joint compared with baseline". Treated target joint bleeds: treated joint bleeds that occurred in a target joint, defined as a joint in which ≥3 treated joint bleeds occurred during the 24 weeks prior to study entry. Treated spontaneous bleeds: treated bleeds with no other known contributing factor such as trauma or procedure/surgery. For all bleed types, bleeds due to surgery/procedure were excluded. Bleeds occurring after dose up-titration have been excluded.
Time Frame: From first dose of emicizumab until dose up-titration or withdrawal from treatment (median [min-max] efficacy period: 103.14 [1.1-108.3] weeks)
Population: Intent-to-Treat (ITT) Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: bleeds per year
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 195
bleeds per year
  Treated Bleeds | 0.5 [0.27 to 0.89]
  All Bleeds | 1.1 [0.80 to 1.47]
  Treated Joint Bleeds | 0.4 [0.15 to 0.86]
  Treated Target Joint Bleeds | 0.2 [0.07 to 0.68]
  Treated Spontaneous Bleeds | 0.3 [0.15 to 0.73]

11. Secondary Outcome: Mean Calculated Annualized Bleed Rates (ABR) for Treated Bleeds, All Bleeds, Treated Joint Bleeds, Treated Target Joint Bleeds, and Treated Spontaneous Bleeds
Description: The number of bleeds over the efficacy period was calculated as: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. Treated bleeds: bleeds followed by a hemophilia medication reported to be a "Treatment for bleed". All bleeds: included both treated and non-treated bleeds. Treated joint bleeds: treated bleeds where bleed type was "joint bleed" accompanied by at least one of following symptoms: "increased swelling or warmth of the skin over the joint", "increasing pain" or "decreased range of motion or difficulty using the joint compared with baseline". Treated target joint bleeds: treated joint bleeds that occurred in a target joint, defined as a joint in which ≥3 treated joint bleeds occurred during the 24 weeks prior to study entry. Treated spontaneous bleeds: treated bleeds with no other known contributing factor such as trauma or procedure/surgery. For all types, bleeds due to surgery/procedure and bleeds occurring after dose up-titration were excluded.
Time Frame: as for outcome 10
Population: Intent-to-Treat (ITT) Population: all enrolled participants
Measure: Mean (95% Confidence Interval); unit: bleeds per year
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 195
bleeds per year
  Treated Bleeds | 0.6 [0.00 to 4.85]
  All Bleeds | 1.3 [0.06 to 6.02]
  Treated Joint Bleeds | 0.4 [0.00 to 4.55]
  Treated Target Joint Bleeds | 0.3 [0.00 to 4.28]
  Treated Spontaneous Bleeds | 0.4 [0.00 to 4.49]

12. Secondary Outcome: Median Calculated Annualized Bleed Rates (ABR) for Treated Bleeds, All Bleeds, Treated Joint Bleeds, Treated Target Joint Bleeds, and Treated Spontaneous Bleeds
Description: as for outcome 11
Time Frame: as for outcome 10
Population: Intent-to-Treat (ITT) Population: all enrolled participants
Measure: Median (Inter-Quartile Range); unit: bleeds per year
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 195
bleeds per year
  Treated Bleeds | 0.0 [0.00 to 0.00]
  All Bleeds | 0.0 [0.00 to 1.01]
  Treated Joint Bleeds | 0.0 [0.00 to 0.00]
  Treated Target Joint Bleeds | 0.0 [0.00 to 0.00]
  Treated Spontaneous Bleeds | 0.0 [0.00 to 0.00]

13. Secondary Outcome: Percentage of Participants by the Categorized Number of Bleeds for Treated Bleeds
Description: Treated bleeds: bleeds followed by a hemophilia medication reported to be a "Treatment for bleed". Bleeds due to surgery/procedure were excluded. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location are counted as one bleed if the second bleed occurs within 72 hours from the last treatment for the first bleed. Included data before up-titration only, for participants whose dose was up-titrated.
Time Frame: as for outcome 10
Population: Intent-to-Treat (ITT) Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 195
Percentage of participants
  0 Bleeds | 82.6 [76.5 to 87.6]
  1-3 Bleeds | 12.3 [8.0 to 17.8]
  4-10 Bleeds | 4.1 [1.8 to 7.9]
  >10 Bleeds | 1.0 [0.1 to 3.7]

14. Secondary Outcome: Percentage of Participants by the Categorized Number of Bleeds for All Bleeds
Description: All bleeds: included both treated and non-treated bleeds. Bleeds due to surgery/procedure were excluded. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location are counted as one bleed if the second bleed occurs within 72 hours from the last treatment for the first bleed. Included data before up-titration only, for participants whose dose was up-titrated.
Time Frame: as for outcome 10
Population: Intent-to-Treat (ITT) Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 195
Percentage of participants
  0 Bleeds | 54.9 [47.6 to 62.0]
  1-3 Bleeds | 30.3 [23.9 to 37.2]
  4-10 Bleeds | 12.3 [8.0 to 17.8]
  >10 Bleeds | 2.6 [0.8 to 5.9]

15. Secondary Outcome: Percentage of Participants by the Categorized Number of Bleeds for Treated Spontaneous Bleeds
Description: Treated spontaneous bleeds: treated bleeds with no other known contributing factor such as trauma or procedure/surgery. Bleeds due to surgery/procedure were excluded. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location are counted as one bleed if the second bleed occurs within 72 hours from the last treatment for the first bleed. Included data before up-titration only, for participants whose dose was up-titrated.
Time Frame: as for outcome 10
Population: Intent-to-Treat (ITT) Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 195
Percentage of participants
  0 Bleeds | 89.2 [84.0 to 93.2]
  1-3 Bleeds | 8.7 [5.2 to 13.6]
  4-10 Bleeds | 1.5 [0.3 to 4.4]
  >10 Bleeds | 0.5 [0.0 to 2.8]

16. Secondary Outcome: Percentage of Participants by the Categorized Calculated Annualized Bleed Rates (ABR) for Treated Bleeds
Description: The number of bleeds over the efficacy period was calculated as an ABR for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. Treated bleeds: bleeds followed by a hemophilia medication reported to be a "Treatment for bleed". Bleeds due to surgery/procedure were excluded. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location are counted as one bleed if the second bleed occurs within 72 hours from the last treatment for the first bleed. Included data before up-titration only, for participants whose dose was up-titrated.
Time Frame: as for outcome 10
Population: Intent-to-Treat (ITT) Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 195
Percentage of participants
  ABR <1 | 90.3 [85.2 to 94.0]
  ABR 1-3.4 | 6.2 [3.2 to 10.5]
  ABR 3.5-10 | 2.6 [0.8 to 5.9]
  ABR >10 | 1.0 [0.1 to 3.7]

17. Secondary Outcome: Percentage of Participants by the Categorized Calculated Annualized Bleed Rates (ABR) for All Bleeds
Description: The number of bleeds over the efficacy period was calculated as an ABR for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. All bleeds: included both treated and non-treated bleeds. Bleeds due to surgery/procedure were excluded. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location are counted as one bleed if the second bleed occurs within 72 hours from the last treatment for the first bleed. Included data before up-titration only, for participants whose dose was up-titrated.
Time Frame: as for outcome 10
Population: Intent-to-Treat (ITT) Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 195
Percentage of participants
  ABR <1 | 72.3 [65.5 to 78.5]
  ABR 1-3.4 | 20.5 [15.1 to 26.9]
  ABR 3.5-10 | 4.6 [2.1 to 8.6]
  ABR >10 | 2.6 [0.8 to 5.9]

18. Secondary Outcome: Percentage of Participants by the Categorized Calculated Annualized Bleed Rates (ABR) for Treated Spontaneous Bleeds
Description: The number of bleeds over the efficacy period was calculated as an ABR for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. Treated spontaneous bleeds: treated bleeds with no other known contributing factor such as trauma or procedure/surgery. Bleeds due to surgery/procedure were excluded. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location are counted as one bleed if the second bleed occurs within 72 hours from the last treatment for the first bleed. Included data before up-titration only, for participants whose dose was up-titrated.
Time Frame: as for outcome 10
Population: Intent-to-Treat (ITT) Population: all enrolled participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 195
Percentage of participants
  ABR <1 | 95.4 [91.4 to 97.9]
  ABR 1-3.4 | 2.6 [0.8 to 5.9]
  ABR 3.5-10 | 1.0 [0.1 to 3.7]
  ABR >10 | 1.0 [0.1 to 3.7]

19. Secondary Outcome: Change From Baseline in the Hemophilia Adult Quality of Life (Haem-A-QoL) Questionnaire Total Score at Specified Timepoints, Adult Participants
Description: The Haem-A-QoL questionnaire was designed for adult participants (greater than or equal to 18 years old) with hemophilia. It consists of 46 items comprising 10 domains: physical health, treatment, work and school, dealing with hemophilia, feelings, familly planning, future, partnerships and sexuality, sports and leisure, and view of yourself. Items are rated by participants with one of five response options: never, seldom, sometimes, often, and always; although, for some items there is also a 'not applicable' option. The Total Score is based on the scores for each domain and ranges from 0 to 100, with lower scores reflective of better quality of life.
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: The number analyzed represents the number of adult participants responding to the questionnaire who had a baseline value and a post-baseline value at a given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 155
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 150
  Baseline (BL) - Value at Visit | 41.09 (16.15)
  Change from BL at Month 3: number analyzed (Participants) | 144
  Change from BL at Month 3 | -17.39 (12.86)
  Change from BL at Month 6: number analyzed (Participants) | 141
  Change from BL at Month 6 | -16.40 (14.58)
  Change from BL at Month 12: number analyzed (Participants) | 140
  Change from BL at Month 12 | -17.44 (14.16)
  Change from BL at Month 18: number analyzed (Participants) | 132
  Change from BL at Month 18 | -16.27 (15.39)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 70
  Change from BL at Early Termination/Study Completion | -14.13 (13.70)
Statistical Analysis 1: Comparison: 1.5 mg/kg Emicizumab QW; Month 3 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 2: Comparison: 1.5 mg/kg Emicizumab QW; Month 6 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 3: Comparison: 1.5 mg/kg Emicizumab QW; Month 12 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 4: Comparison: 1.5 mg/kg Emicizumab QW; Month 18 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 5: Comparison: 1.5 mg/kg Emicizumab QW; Early Terminatinon/Study Completion vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test

20. Secondary Outcome: Percentage of Participants With an Improvement From Baseline Greater Than the Responder Threshold for the Hemophilia Adult Quality of Life (Haem-A-QoL) Questionnaire Total Score at Specified Timepoints
Description: The Haem-A-QoL questionnaire was designed for adult participants (greater than or equal to 18 years old) with hemophilia. It consists of 46 items comprising 10 domains: physical health, treatment, work and school, dealing with hemophilia, feelings, familly planning, future, partnerships and sexuality, sports and leisure, and view of yourself. Items are rated by participants with one of five response options: never, seldom, sometimes, often, and always; although, for some items there is also a 'not applicable' option. The Total Score is based on the scores for each domain and ranges from 0 to 100, with lower scores reflective of better quality of life. An improvement larger than the responder threshold was defined as a decrease from baseline of at least 7 points in the Haem-A-QoL Total score.
Time Frame: At 3, 6, 12, and 18 months
Population: The number analyzed represents the number of adult participants responding to the questionnaire who had a post-baseline value at a given timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 155
Percentage of participants
  Month 3: number analyzed (Participants) | 147
  Month 3 | 78.2
  Month 6: number analyzed (Participants) | 145
  Month 6 | 72.4
  Month 12: number analyzed (Participants) | 144
  Month 12 | 70.8
  Month 18: number analyzed (Participants) | 136
  Month 18 | 69.9

21. Secondary Outcome: Change From Baseline in the Hemophilia Adult Quality of Life (Haem-A-QoL) Questionnaire Physical Health Domain Score at Specified Timepoints, Adult Participants
Description: The Haem-A-QoL questionnaire was designed for adult participants (greater than or equal to 18 years old) with hemophilia. It consists of 46 items comprising 10 domains: physical health, treatment, work and school, dealing with hemophilia, feelings, familly planning, future, partnerships and sexuality, sports and leisure, and view of yourself. Items are rated by participants with one of five response options: never, seldom, sometimes, often, and always; although, for some items there is also a 'not applicable' option. Scale scores for each domain range from 0 to 100, with lower scores reflective of better quality of life.
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 155
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 150
  Baseline (BL) - Value at Visit | 51.13 (23.02)
  Change from BL at Month 3: number analyzed (Participants) | 144
  Change from BL at Month 3 | -27.36 (20.70)
  Change from BL at Month 6: number analyzed (Participants) | 141
  Change from BL at Month 6 | -26.10 (23.12)
  Change from BL at Month 12: number analyzed (Participants) | 140
  Change from BL at Month 12 | -25.21 (23.31)
  Change from BL at Month 18: number analyzed (Participants) | 132
  Change from BL at Month 18 | -23.14 (24.51)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 70
  Change from BL at Early Termination/Study Completion | -23.29 (25.16)
Statistical Analysis 1: Comparison: 1.5 mg/kg Emicizumab QW; Month 3 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 2: Comparison: 1.5 mg/kg Emicizumab QW; Month 6 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 3: Comparison: 1.5 mg/kg Emicizumab QW; Month 12 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 4: Comparison: 1.5 mg/kg Emicizumab QW; Month 18 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 5: Comparison: 1.5 mg/kg Emicizumab QW; Early Terminatinon/Study Completion vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test

22. Secondary Outcome: Percentage of Participants With an Improvement From Baseline Greater Than the Responder Threshold for the Hemophilia Adult Quality of Life (Haem-A-QoL) Questionnaire Physical Health Domain Score at Specified Timepoints
Description: The Haem-A-QoL questionnaire was designed for adult participants (greater than or equal to 18 years old) with hemophilia. It consists of 46 items comprising 10 domains: physical health, treatment, work and school, dealing with hemophilia, feelings, familly planning, future, partnerships and sexuality, sports and leisure, and view of yourself. Items are rated by participants with one of five response options: never, seldom, sometimes, often, and always; although, for some items there is also a 'not applicable' option. Scale scores for each domain range from 0 to 100, with lower scores reflective of better quality of life. An improvement larger than the responder threshold was defined as a decrease from baseline of at least 10 points in the Haem-A-QoL Physical Health domain score.
Time Frame: At 3, 6, 12, and 18 months
Population: as for outcome 20
Measure: Number; unit: Percentage of participants
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 155
Percentage of participants
  Month 3: number analyzed (Participants) | 147
  Month 3 | 79.6
  Month 6: number analyzed (Participants) | 145
  Month 6 | 74.5
  Month 12: number analyzed (Participants) | 144
  Month 12 | 72.9
  Month 18: number analyzed (Participants) | 136
  Month 18 | 71.3

23. Secondary Outcome: Change From Baseline in the Hemophilia Adult Quality of Life (Haem-A-QoL) Questionnaire Treatment Domain Score at Specified Timepoints, Adult Participants
Description: as for outcome 21
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 155
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 150
  Baseline (BL) - Value at Visit | 39.40 (19.89)
  Change from BL at Month 3: number analyzed (Participants) | 144
  Change from BL at Month 3 | -23.44 (22.07)
  Change from BL at Month 6: number analyzed (Participants) | 141
  Change from BL at Month 6 | -21.01 (23.74)
  Change from BL at Month 12: number analyzed (Participants) | 140
  Change from BL at Month 12 | -22.21 (22.57)
  Change from BL at Month 18: number analyzed (Participants) | 132
  Change from BL at Month 18 | -20.34 (25.37)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 70
  Change from BL at Early Termination/Study Completion | -21.16 (22.31)

24. Secondary Outcome: Change From Baseline in the Hemophilia Adult Quality of Life (Haem-A-QoL) Questionnaire Work and School Domain Score at Specified Timepoints, Adult Participants
Description: as for outcome 21
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 155
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 125
  Baseline (BL) - Value at Visit | 39.23 (25.31)
  Change from BL at Month 3: number analyzed (Participants) | 114
  Change from BL at Month 3 | -21.40 (26.51)
  Change from BL at Month 6: number analyzed (Participants) | 106
  Change from BL at Month 6 | -21.91 (27.17)
  Change from BL at Month 12: number analyzed (Participants) | 106
  Change from BL at Month 12 | -22.43 (25.55)
  Change from BL at Month 18: number analyzed (Participants) | 101
  Change from BL at Month 18 | -21.43 (26.65)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 51
  Change from BL at Early Termination/Study Completion | -18.83 (29.54)

25. Secondary Outcome: Change From Baseline in the Hemophilia Adult Quality of Life (Haem-A-QoL) Questionnaire Dealing With Hemophilia Domain Score at Specified Timepoints, Adult Participants
Description: as for outcome 21
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 155
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 150
  Baseline (BL) - Value at Visit | 26.61 (19.76)
  Change from BL at Month 3: number analyzed (Participants) | 144
  Change from BL at Month 3 | 5.32 (30.06)
  Change from BL at Month 6: number analyzed (Participants) | 141
  Change from BL at Month 6 | 5.73 (28.14)
  Change from BL at Month 12: number analyzed (Participants) | 140
  Change from BL at Month 12 | 5.24 (29.18)
  Change from BL at Month 18: number analyzed (Participants) | 132
  Change from BL at Month 18 | 7.70 (29.75)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 70
  Change from BL at Early Termination/Study Completion | 10.60 (33.42)

26. Secondary Outcome: Change From Baseline in the Hemophilia Adult Quality of Life (Haem-A-QoL) Questionnaire Feelings Domain Score at Specified Timepoints, Adult Participants
Description: as for outcome 21
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 155
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 150
  Baseline (BL) - Value at Visit | 36.25 (24.53)
  Change from BL at Month 3: number analyzed (Participants) | 144
  Change from BL at Month 3 | -21.22 (22.69)
  Change from BL at Month 6: number analyzed (Participants) | 141
  Change from BL at Month 6 | -20.88 (24.11)
  Change from BL at Month 12: number analyzed (Participants) | 140
  Change from BL at Month 12 | -22.37 (23.78)
  Change from BL at Month 18: number analyzed (Participants) | 132
  Change from BL at Month 18 | -19.55 (25.43)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 70
  Change from BL at Early Termination/Study Completion | -17.95 (23.62)

27. Secondary Outcome: Change From Baseline in the Hemophilia Adult Quality of Life (Haem-A-QoL) Questionnaire Family Planning Domain Score at Specified Timepoints, Adult Participants
Description: as for outcome 21
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 155
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 91
  Baseline (BL) - Value at Visit | 25.64 (28.49)
  Change from BL at Month 3: number analyzed (Participants) | 67
  Change from BL at Month 3 | -8.64 (20.95)
  Change from BL at Month 6: number analyzed (Participants) | 68
  Change from BL at Month 6 | -9.07 (20.78)
  Change from BL at Month 12: number analyzed (Participants) | 65
  Change from BL at Month 12 | -10.83 (22.51)
  Change from BL at Month 18: number analyzed (Participants) | 58
  Change from BL at Month 18 | -12.39 (25.20)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 26
  Change from BL at Early Termination/Study Completion | -9.38 (24.81)

28. Secondary Outcome: Change From Baseline in the Hemophilia Adult Quality of Life (Haem-A-QoL) Questionnaire Future Domain Score at Specified Timepoints, Adult Participants
Description: as for outcome 21
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 155
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 150
  Baseline (BL) - Value at Visit | 42.70 (21.95)
  Change from BL at Month 3: number analyzed (Participants) | 144
  Change from BL at Month 3 | -15.56 (17.63)
  Change from BL at Month 6: number analyzed (Participants) | 141
  Change from BL at Month 6 | -15.46 (17.83)
  Change from BL at Month 12: number analyzed (Participants) | 140
  Change from BL at Month 12 | -14.46 (20.10)
  Change from BL at Month 18: number analyzed (Participants) | 132
  Change from BL at Month 18 | -14.43 (19.83)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 70
  Change from BL at Early Termination/Study Completion | -13.29 (19.56)

29. Secondary Outcome: Change From Baseline in the Hemophilia Adult Quality of Life (Haem-A-QoL) Questionnaire Partnership and Sexuality Domain Score at Specified Timepoints, Adult Participants
Description: as for outcome 21
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 155
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 150
  Baseline (BL) - Value at Visit | 23.17 (28.65)
  Change from BL at Month 3: number analyzed (Participants) | 144
  Change from BL at Month 3 | -7.35 (25.25)
  Change from BL at Month 6: number analyzed (Participants) | 141
  Change from BL at Month 6 | -6.03 (22.76)
  Change from BL at Month 12: number analyzed (Participants) | 140
  Change from BL at Month 12 | -7.74 (27.60)
  Change from BL at Month 18: number analyzed (Participants) | 132
  Change from BL at Month 18 | -9.72 (28.16)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 70
  Change from BL at Early Termination/Study Completion | -4.05 (21.32)

30. Secondary Outcome: Change From Baseline in the Hemophilia Adult Quality of Life (Haem-A-QoL) Questionnaire Sports and Leisure Domain Score at Specified Timepoints, Adult Participants
Description: as for outcome 21
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 155
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 114
  Baseline (BL) - Value at Visit | 68.86 (21.24)
  Change from BL at Month 3: number analyzed (Participants) | 89
  Change from BL at Month 3 | -19.65 (23.67)
  Change from BL at Month 6: number analyzed (Participants) | 83
  Change from BL at Month 6 | -17.63 (25.86)
  Change from BL at Month 12: number analyzed (Participants) | 87
  Change from BL at Month 12 | -22.56 (22.17)
  Change from BL at Month 18: number analyzed (Participants) | 76
  Change from BL at Month 18 | -20.20 (25.86)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 42
  Change from BL at Early Termination/Study Completion | -20.65 (28.65)

31. Secondary Outcome: Change From Baseline in the Hemophilia Adult Quality of Life (Haem-A-QoL) Questionnaire View of Yourself Domain Score at Specified Timepoints, Adult Participants
Description: as for outcome 21
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 155
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 150
  Baseline (BL) - Value at Visit | 43.57 (22.05)
  Change from BL at Month 3: number analyzed (Participants) | 144
  Change from BL at Month 3 | -13.51 (20.63)
  Change from BL at Month 6: number analyzed (Participants) | 141
  Change from BL at Month 6 | -15.04 (21.19)
  Change from BL at Month 12: number analyzed (Participants) | 140
  Change from BL at Month 12 | -15.71 (19.88)
  Change from BL at Month 18: number analyzed (Participants) | 132
  Change from BL at Month 18 | -15.19 (21.88)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 70
  Change from BL at Early Termination/Study Completion | -9.50 (20.70)

32. Secondary Outcome: Change From Baseline in the Hemophilia Quality of Life Short Form (Haemo-QoL-SF) Questionnaire Total Score at Specified Timepoints, Adolescent Participants
Description: The Haemo-QoL-SF was designed as a series of age-related questionnaires to measure health-related quality of life in children and adolescents (12-17 year olds) with hemophilia. This version contains 35 items and covers nine domains considered relevant for children's health-related quality of life: physical health, treatment, sports and school, dealing with hemophilia, feelings, family, friends, other people, and view of yourself. Items are rated by participants with one of five response options: never, seldom, sometimes, often, and always. The Total Score is derived from the scores for all domains and scale scores range from 0 to 100, with a lower score reflective of better health-related quality of life.
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: The number analyzed represents the number of adolescent participants responding to the questionnaire who had a baseline value and a post-baseline value at a given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 40
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 35
  Baseline (BL) - Value at Visit | 35.10 (12.42)
  Change from BL at Month 3: number analyzed (Participants) | 32
  Change from BL at Month 3 | -9.60 (12.51)
  Change from BL at Month 6: number analyzed (Participants) | 34
  Change from BL at Month 6 | -12.65 (12.72)
  Change from BL at Month 12: number analyzed (Participants) | 32
  Change from BL at Month 12 | -13.57 (13.20)
  Change from BL at Month 18: number analyzed (Participants) | 35
  Change from BL at Month 18 | -14.02 (11.83)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 18
  Change from BL at Early Termination/Study Completion | -18.37 (17.53)
Statistical Analysis 1: Comparison: 1.5 mg/kg Emicizumab QW; Month 3 vs. Baseline; Test type: Superiority; p = 0.0001, Paired t-test
Statistical Analysis 2: Comparison: 1.5 mg/kg Emicizumab QW; Month 6 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 3: Comparison: 1.5 mg/kg Emicizumab QW; Month 12 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 4: Comparison: 1.5 mg/kg Emicizumab QW; Month 18 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 5: Comparison: 1.5 mg/kg Emicizumab QW; Early Terminatinon/Study Completion vs. Baseline; Test type: Superiority; p = 0.0004, Paired t-test

33. Secondary Outcome: Percentage of Participants With an Improvement From Baseline Greater Than the Responder Threshold for the Hemophilia Quality of Life Short Form (Haemo-QoL-SF) Questionnaire Total Score at Specified Timepoints
Description: The Haemo-QoL-SF was designed as a series of age-related questionnaires to measure health-related quality of life in children and adolescents (12-17 year olds) with hemophilia. This version contains 35 items and covers nine domains considered relevant for children's health-related quality of life: physical health, treatment, sports and school, dealing with hemophilia, feelings, family, friends, other people, and view of yourself. Items are rated by participants with one of five response options: never, seldom, sometimes, often, and always. The Total Score is derived from the scores for all domains and scale scores range from 0 to 100, with a lower score reflective of better health-related quality of life. An improvement larger than the responder threshold was defined as a decrease of at least 5 points in the Haemo-QoL-SF Total score.
Time Frame: At 3, 6, 12, and 18 months
Population: The number analyzed represents the number of adolescent participants responding to the questionnaire who had a post-baseline value at a given timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 40
Percentage of participants
  Month 3: number analyzed (Participants) | 36
  Month 3 | 63.9
  Month 6: number analyzed (Participants) | 37
  Month 6 | 75.7
  Month 12: number analyzed (Participants) | 36
  Month 12 | 75.0
  Month 18: number analyzed (Participants) | 39
  Month 18 | 69.2

34. Secondary Outcome: Change From Baseline in the Hemophilia Quality of Life Short Form (Haemo-QoL-SF) Questionnaire Physical Health Domain Score at Specified Timepoints, Adolescent Participants
Description: The Haemo-QoL-SF was designed as a series of age-related questionnaires to measure health-related quality of life in children and adolescents (12-17 year olds) with hemophilia. This version contains 35 items and covers nine domains considered relevant for children's health-related quality of life: physical health, treatment, sports and school, dealing with hemophilia, feelings, family, friends, other people, and view of yourself. Items are rated by participants with one of five response options: never, seldom, sometimes, often, and always. Scale scores range from 0 to 100, with a lower score reflective of better health-related quality of life.
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 40
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 35
  Baseline (BL) - Value at Visit | 42.14 (18.40)
  Change from BL at Month 3: number analyzed (Participants) | 32
  Change from BL at Month 3 | -29.10 (20.12)
  Change from BL at Month 6: number analyzed (Participants) | 34
  Change from BL at Month 6 | -29.78 (17.55)
  Change from BL at Month 12: number analyzed (Participants) | 32
  Change from BL at Month 12 | -30.47 (20.74)
  Change from BL at Month 18: number analyzed (Participants) | 35
  Change from BL at Month 18 | -30.71 (18.83)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 18
  Change from BL at Early Termination/Study Completion | -34.03 (25.66)
Statistical Analysis 1: Comparison: 1.5 mg/kg Emicizumab QW; Month 3 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 2: Comparison: 1.5 mg/kg Emicizumab QW; Month 6 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 3: Comparison: 1.5 mg/kg Emicizumab QW; Month 12 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 4: Comparison: 1.5 mg/kg Emicizumab QW; Month 18 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 5: Comparison: 1.5 mg/kg Emicizumab QW; Early Terminatinon/Study Completion vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test

35. Secondary Outcome: Percentage of Participants With an Improvement From Baseline Greater Than the Responder Threshold for the Hemophilia Quality of Life Short Form (Haemo-QoL-SF) Questionnaire Physical Health Domain Score at Specified Timepoints
Description: The Haemo-QoL-SF was designed as a series of age-related questionnaires to measure health-related quality of life in children and adolescents (12-17 year olds) with hemophilia. This version contains 35 items and covers nine domains considered relevant for children's health-related quality of life: physical health, treatment, sports and school, dealing with hemophilia, feelings, family, friends, other people, and view of yourself. Items are rated by participants with one of five response options: never, seldom, sometimes, often, and always. Scale scores range from 0 to 100, with a lower score reflective of better health-related quality of life. An improvement larger than the responder threshold was defined as a decrease of at least 10 points in the Haemo-QoL-SF Physical Health domain score.
Time Frame: At 3, 6, 12, and 18 months
Population: as for outcome 33
Measure: Number; unit: Percentage of participants
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 40
Percentage of participants
  Month 3: number analyzed (Participants) | 36
  Month 3 | 77.8
  Month 6: number analyzed (Participants) | 37
  Month 6 | 78.4
  Month 12: number analyzed (Participants) | 36
  Month 12 | 75.0
  Month 18: number analyzed (Participants) | 39
  Month 18 | 79.5

36. Secondary Outcome: Change From Baseline in the Hemophilia Quality of Life Short Form (Haemo-QoL-SF) Questionnaire Treatment Domain Score at Specified Timepoints, Adolescent Participants
Description: as for outcome 34
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 40
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 35
  Baseline (BL) - Value at Visit | 31.61 (18.12)
  Change from BL at Month 3: number analyzed (Participants) | 32
  Change from BL at Month 3 | -9.38 (20.94)
  Change from BL at Month 6: number analyzed (Participants) | 34
  Change from BL at Month 6 | -8.64 (23.23)
  Change from BL at Month 12: number analyzed (Participants) | 32
  Change from BL at Month 12 | -10.74 (21.31)
  Change from BL at Month 18: number analyzed (Participants) | 35
  Change from BL at Month 18 | -12.68 (21.68)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 18
  Change from BL at Early Termination/Study Completion | -20.83 (23.87)

37. Secondary Outcome: Change From Baseline in the Hemophilia Quality of Life Short Form (Haemo-QoL-SF) Questionnaire Sports and School Domain Score at Specified Timepoints, Adolescent Participants
Description: as for outcome 34
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 40
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 35
  Baseline (BL) - Value at Visit | 62.32 (21.30)
  Change from BL at Month 3: number analyzed (Participants) | 32
  Change from BL at Month 3 | -15.82 (25.55)
  Change from BL at Month 6: number analyzed (Participants) | 34
  Change from BL at Month 6 | -20.04 (29.27)
  Change from BL at Month 12: number analyzed (Participants) | 32
  Change from BL at Month 12 | -22.07 (26.71)
  Change from BL at Month 18: number analyzed (Participants) | 35
  Change from BL at Month 18 | -28.21 (27.80)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 18
  Change from BL at Early Termination/Study Completion | -23.61 (28.16)

38. Secondary Outcome: Change From Baseline in the Hemophilia Quality of Life Short Form (Haemo-QoL-SF) Questionnaire Dealing With Hemophilia Domain Score at Specified Timepoints, Adolescent Participants
Description: as for outcome 34
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 40
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 35
  Baseline (BL) - Value at Visit | 24.11 (14.79)
  Change from BL at Month 3: number analyzed (Participants) | 32
  Change from BL at Month 3 | -7.23 (18.25)
  Change from BL at Month 6: number analyzed (Participants) | 34
  Change from BL at Month 6 | -7.72 (17.75)
  Change from BL at Month 12: number analyzed (Participants) | 32
  Change from BL at Month 12 | -10.35 (20.24)
  Change from BL at Month 18: number analyzed (Participants) | 35
  Change from BL at Month 18 | -3.39 (25.70)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 18
  Change from BL at Early Termination/Study Completion | -12.50 (23.48)

39. Secondary Outcome: Change From Baseline in the Hemophilia Quality of Life Short Form (Haemo-QoL-SF) Questionnaire Feelings Domain Score at Specified Timepoints, Adolescent Participants
Description: as for outcome 34
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 40
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 35
  Baseline (BL) - Value at Visit | 26.43 (25.10)
  Change from BL at Month 3: number analyzed (Participants) | 32
  Change from BL at Month 3 | -9.57 (20.08)
  Change from BL at Month 6: number analyzed (Participants) | 34
  Change from BL at Month 6 | -16.36 (21.54)
  Change from BL at Month 12: number analyzed (Participants) | 32
  Change from BL at Month 12 | -13.09 (22.80)
  Change from BL at Month 18: number analyzed (Participants) | 35
  Change from BL at Month 18 | -15.18 (25.51)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 18
  Change from BL at Early Termination/Study Completion | -23.96 (32.67)

40. Secondary Outcome: Change From Baseline in the Hemophilia Quality of Life Short Form (Haemo-QoL-SF) Questionnaire Family Domain Score at Specified Timepoints, Adolescent Participants
Description: as for outcome 34
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 40
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 35
  Baseline (BL) - Value at Visit | 46.07 (20.79)
  Change from BL at Month 3: number analyzed (Participants) | 32
  Change from BL at Month 3 | -6.84 (15.66)
  Change from BL at Month 6: number analyzed (Participants) | 34
  Change from BL at Month 6 | -11.95 (20.84)
  Change from BL at Month 12: number analyzed (Participants) | 32
  Change from BL at Month 12 | -14.84 (23.32)
  Change from BL at Month 18: number analyzed (Participants) | 35
  Change from BL at Month 18 | -15.36 (21.67)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 18
  Change from BL at Early Termination/Study Completion | -15.28 (19.08)

41. Secondary Outcome: Change From Baseline in the Hemophilia Quality of Life Short Form (Haemo-QoL-SF) Questionnaire Friends Domain Score at Specified Timepoints, Adolescent Participants
Description: as for outcome 34
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 40
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 35
  Baseline (BL) - Value at Visit | 35.95 (26.02)
  Change from BL at Month 3: number analyzed (Participants) | 32
  Change from BL at Month 3 | -0.52 (24.95)
  Change from BL at Month 6: number analyzed (Participants) | 34
  Change from BL at Month 6 | -3.19 (28.13)
  Change from BL at Month 12: number analyzed (Participants) | 32
  Change from BL at Month 12 | -5.47 (27.57)
  Change from BL at Month 18: number analyzed (Participants) | 35
  Change from BL at Month 18 | -5.95 (36.41)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 18
  Change from BL at Early Termination/Study Completion | -7.41 (31.56)

42. Secondary Outcome: Change From Baseline in the Hemophilia Quality of Life Short Form (Haemo-QoL-SF) Questionnaire Other People Domain Score at Specified Timepoints, Adolescent Participants
Description: as for outcome 34
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 40
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 35
  Baseline (BL) - Value at Visit | 21.43 (17.50)
  Change from BL at Month 3: number analyzed (Participants) | 32
  Change from BL at Month 3 | -2.93 (18.72)
  Change from BL at Month 6: number analyzed (Participants) | 34
  Change from BL at Month 6 | -5.51 (19.08)
  Change from BL at Month 12: number analyzed (Participants) | 32
  Change from BL at Month 12 | -8.01 (18.53)
  Change from BL at Month 18: number analyzed (Participants) | 35
  Change from BL at Month 18 | -6.79 (17.51)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 18
  Change from BL at Early Termination/Study Completion | -11.81 (18.55)

43. Secondary Outcome: Change From Baseline in the Hemophilia Quality of Life Short Form (Haemo-QoL-SF) Questionnaire View of Yourself Domain Score at Specified Timepoints, Adolescent Participants
Description: as for outcome 34
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 40
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 35
  Baseline (BL) - Value at Visit | 26.07 (22.04)
  Change from BL at Month 3: number analyzed (Participants) | 32
  Change from BL at Month 3 | -2.73 (26.03)
  Change from BL at Month 6: number analyzed (Participants) | 34
  Change from BL at Month 6 | -8.27 (23.27)
  Change from BL at Month 12: number analyzed (Participants) | 32
  Change from BL at Month 12 | -5.08 (24.82)
  Change from BL at Month 18: number analyzed (Participants) | 35
  Change from BL at Month 18 | -5.89 (21.54)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 18
  Change from BL at Early Termination/Study Completion | -13.19 (26.59)

44. Secondary Outcome: Change From Baseline in the EuroQoL Five-Dimension-Five Levels Questionnaire (EQ-5D-5L) Index Utility Score at Specified Timepoints
Description: The EQ-5D-5L is a generic, self-reported, preference-based health utility measure that consists of six questions and is used to assess health status and inform pharmacoeconomic evaluations. The index utility score is based on the participant's assessment of their health on five scales: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It ranges from -0.224 to 1, with 0 corresponding to death and 1 corresponding to full health; negative values correspond to health states worse than death. Higher scores indicate better quality of life.
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: The number analyzed represents the number of participants responding to the questionnaire who had a baseline value and a post-baseline value at a given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 195
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 188
  Baseline (BL) - Value at Visit | 0.67 (0.23)
  Change from BL at Month 3: number analyzed (Participants) | 182
  Change from BL at Month 3 | 0.08 (0.18)
  Change from BL at Month 6: number analyzed (Participants) | 178
  Change from BL at Month 6 | 0.11 (0.18)
  Change from BL at Month 12: number analyzed (Participants) | 176
  Change from BL at Month 12 | 0.09 (0.19)
  Change from BL at Month 18: number analyzed (Participants) | 170
  Change from BL at Month 18 | 0.07 (0.21)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 89
  Change from BL at Early Termination/Study Completion | 0.10 (0.22)
Statistical Analysis 1: Comparison: 1.5 mg/kg Emicizumab QW; Month 3 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 2: Comparison: 1.5 mg/kg Emicizumab QW; Month 6 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 3: Comparison: 1.5 mg/kg Emicizumab QW; Month 12 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 4: Comparison: 1.5 mg/kg Emicizumab QW; Month 18 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 5: Comparison: 1.5 mg/kg Emicizumab QW; Early Terminatinon/Study Completion vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test

45. Secondary Outcome: Change From Baseline in the EuroQoL Five-Dimension-Five Levels Questionnaire (EQ-5D-5L) Quality-of-Life Visual Analogue Scale (VAS) Score at Specified Timepoints
Description: The EQ-5D-5L is a generic, self-reported, preference-based health utility measure that consists of six questions and is used to assess health status and inform pharmacoeconomic evaluations. The visual analogue scale (VAS) ranges from 0 to 100 points, on which the participant self-assesses their current health status; 0 being the worst health you can imagine and 100 being the best health you can imagine. Higher scores are reflective of better health.
Time Frame: Baseline (Week 1), 3, 6, 12, and 18 months, and at Early Termination or Study Completion (up to 24 months)
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 195
score on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 188
  Baseline (BL) - Value at Visit | 71.01 (19.41)
  Change from BL at Month 3: number analyzed (Participants) | 182
  Change from BL at Month 3 | 8.02 (18.70)
  Change from BL at Month 6: number analyzed (Participants) | 177
  Change from BL at Month 6 | 10.27 (17.24)
  Change from BL at Month 12: number analyzed (Participants) | 176
  Change from BL at Month 12 | 10.69 (18.18)
  Change from BL at Month 18: number analyzed (Participants) | 170
  Change from BL at Month 18 | 9.49 (21.08)
  Change from BL at Early Termination/Study Completion: number analyzed (Participants) | 89
  Change from BL at Early Termination/Study Completion | 14.52 (17.91)
Statistical Analysis 1: Comparison: 1.5 mg/kg Emicizumab QW; Month 3 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 2: Comparison: 1.5 mg/kg Emicizumab QW; Month 6 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 3: Comparison: 1.5 mg/kg Emicizumab QW; Month 12 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 4: Comparison: 1.5 mg/kg Emicizumab QW; Month 18 vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test
Statistical Analysis 5: Comparison: 1.5 mg/kg Emicizumab QW; Early Terminatinon/Study Completion vs. Baseline; Test type: Superiority; p < 0.0001, Paired t-test

46. Secondary Outcome: Percentage of Participants Who Preferred the New Emicizumab Treatment or the Old Hemophilia Treatment, or Without Treatment Preference, as Assessed by the EmiPref Questionnaire
Description: The EmiPref questionnaire asked participants to specify the treatment they would prefer to continue to receive after receiving treatment with their previous episodic or prophylactic regimen and subcutaneous (SC) emicizumab, or if they had no preference. The 95% confidence intervals were calculated for one sample binomial using the Pearson-Clopper method.
Time Frame: Month 3
Population: The number of participants analyzed represents the total number who responded to this questionnaire.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 179
Percentage of participants
  Prefer the New Study Drug Treatment (Emicizumab) | 96.6 [92.85 to 98.76]
  Prefer my Old Hemophilia Treatment | 0.6 [0.01 to 3.07]
  Have no Preference | 2.8 [0.91 to 6.40]

47. Secondary Outcome: Number and Percentage of Participants With Anti-Drug Antibodies (ADAs) Against Emicizumab at Anytime Post-Baseline
Description: 'Total ADA Negative' is the sum of all subjects who tested negative for ADA in the 2 following categories: 'ADA Negative', those who are pre-dose ADA negative or are missing pre-dose ADA data and who have all negative post-dose ADA results; and 'ADA Negative (Treatment Unaffected)', a subset who are pre-dose ADA positive but do not have a ≥4-fold increase in post-dose ADA levels compared to baseline measurement. 'Total ADA Positive' is the sum of all subjects who tested positive for ADA in the 2 following categories: 'ADA Positive (Treatment Boosted)', those who are pre-dose ADA positive and have a ≥4-fold increase in post-dose ADA levels compared to baseline measurement; and 'ADA Positive (Treatment Induced)', those who are pre-dose ADA negative or missing data and who have at least one post-dose ADA positive sample.
Time Frame: Baseline (Week 1), Week 5, and at 3, 6, 9, 12, and 18 months, and at early termination/study completion (up to 24 months)
Population: Safety Population: all participants who received at least one dose of emicizumab. The number analyzed included participants with at least one baseline and one post-baseline assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 193
Participants
  Total ADA Negative (Neg + Neg Unaffected) | 183
  ADA Negative | 180
  ADA Negative (Treatment Unaffected) | 3
  Total ADA Positive (Boosted + Induced) | 10
  ADA Positive (Treatment Boosted) | 2
  ADA Positive (Treatment Induced) | 8

48. Secondary Outcome: Mean Trough Plasma Concentrations of Emicizumab at Specified Timepoints
Description: The trough concentration is a measure of the plasma concentration of a study drug at the end of of the dosage interval.
Time Frame: Pre-dose at Weeks 2, 3, and 5, Months 3, 6, 12, and 18, and at treatment discontinuation (up to 2 years)
Population: Pharmacokinetic-Evaluable Population: all participants who received at least one dose of emicizumab and had at least one post-baseline emicizumab concentration result.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (μg/mL)
Arm/Group | 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 193
micrograms per millilitre (μg/mL)
  Week 2: number analyzed (Participants) | 188
  Week 2 | 16.7 (5.5)
  Week 3: number analyzed (Participants) | 190
  Week 3 | 30.7 (9.2)
  Week 5: number analyzed (Participants) | 187
  Week 5 | 52.4 (15.5)
  Month 3: number analyzed (Participants) | 186
  Month 3 | 52.5 (18.3)
  Month 6: number analyzed (Participants) | 183
  Month 6 | 53.4 (19.3)
  Month 12: number analyzed (Participants) | 183
  Month 12 | 54.2 (20.6)
  Month 18: number analyzed (Participants) | 171
  Month 18 | 53.6 (18.3)
  Treatment Discontinuation: number analyzed (Participants) | 154
  Treatment Discontinuation | 54.6 (19.0)

ADVERSE EVENTS:
Time Frame: From Baseline until study completion (up to 2 years)
Arm/Group | 1.5 mg/kg Emicizumab QW
All-Cause Mortality (participants affected / at risk) | 2/193
Serious Adverse Events (participants affected / at risk) | 31/193
Other Adverse Events (participants affected / at risk) | 104/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 mg/kg Emicizumab QW (N=193)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
ABDOMINAL COMPARTMENT SYNDROME (Gastrointestinal disorders) | 1 (1)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (5)
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 1 (1)
SUBCAPSULAR HEPATIC HAEMATOMA (Hepatobiliary disorders) | 1 (1)
ABSCESS (Infections and infestations) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1)
CATHETER SITE ABSCESS (Infections and infestations) | 2 (2)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1)
INFECTED SKIN ULCER (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
WOUND INFECTION (Infections and infestations) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
INJURY (Injury, poisoning and procedural complications) | 1 (1)
JOINT INJURY (Injury, poisoning and procedural complications) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 2 (2)
WOUND HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1)
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
HAEMATOMA MUSCLE (Musculoskeletal and connective tissue disorders) | 2 (2)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 1 (1)
TENSION HEADACHE (Nervous system disorders) | 1 (1)
DEVICE DISLOCATION (Product Issues) | 1 (1)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 (1)
RENAL PAIN (Renal and urinary disorders) | 1 (1)
URETEROLITHIASIS (Renal and urinary disorders) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CENTRAL VENOUS CATHETER REMOVAL (Surgical and medical procedures) | 1 (1)
HAEMATOMA (Vascular disorders) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 mg/kg Emicizumab QW (N=193)
INJECTION SITE REACTION (General disorders) | 22 (29)
PYREXIA (General disorders) | 21 (26)
INFLUENZA (Infections and infestations) | 16 (25)
NASOPHARYNGITIS (Infections and infestations) | 30 (47)
FALL (Injury, poisoning and procedural complications) | 12 (16)
LIMB INJURY (Injury, poisoning and procedural complications) | 10 (12)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 33 (52)
HEADACHE (Nervous system disorders) | 29 (52)
COUGH (Respiratory, thoracic and mediastinal disorders) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT03191799/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT03191799/SAP_001.pdf